CLINICAL TRIAL: NCT04150874
Title: Contrast-Enhanced Ultrasound for the Evaluation of Changes in Tumor Blood Flow and the Surrounding Hepatic Parenchyma Before, During and After Hepatic Artery Embolization
Brief Title: Contrast-Enhanced Ultrasound for the Evaluation of Changes in Tumor Blood Flow Surrounding HAE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-19974
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Hepatic Artery Embolization; Liver Metastases; Radioembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lumason Microbubbles (Experimental): Participants will receive an IV administrative of Lumason® microbubbles, prior to radioembolization. 2 doses of 2.5mL will be administered
  Interventions: Diagnostic Test: Lumason®

INTERVENTIONS:
Diagnostic Test: Lumason® — Hepatic artery embolization using standard of care radioembolization and assessment of tumor and hepatic parenchymal perfusion kinetics before, during and after treatment with standard of care iodinated contrast (at the time of Y90 radioembolization treatment) and standard of care follow-up with multiphase CT or MRI with the addition of study agent Lumason microbubbles for contrast-enhanced ultrasound (which will be performed concurrently with standard evaluation).

SUMMARY:
The purpose of the study is to find out if a study agent called Lumason® microbubbles may be helpful for people with lesions in the liver. It is possible it may help determine an early response to radioembolization and/or help demonstrate radiation toxicity to the surrounding liver.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Men and women >18 years of age.
* Histologically or cytologically confirmed hepatocellular carcinoma or meet imaging criteria for a diagnosis of hepatocellular carcinoma with tumor burden dominant in the liver.
* Participants must have measurable disease, by CT or MRI per mRECIST, not be a candidate for surgical resection based on unresectability, anatomy, anesthesia risk, patient preference.
* Serum Bilirubin ≤ 2.0
* Platelet count > 50,000/ul (corrected if needed)
* INR ≤ 1.5 (corrected if needed) 9. Serum creatinine < 2.0 mg/dl

Exclusion Criteria:

* Participants must be at least one month beyond prior chemotherapy, ablation or surgery, and have recovered from all therapy-associated toxicities.
* History of severe allergic reaction to intravenous contrast media (iodinated and gadoliniumbased) or any agents used during the embolization; participant cannot be medicated against allergic reaction prior to embolization or contrast enhanced ultrasound.
* History of hypersensitivity reactions to sulfur hexafluoride lipid microsphere components or to any of the inactive ingredients in Lumason® microbubbles
* Active infection
* Participants with unstable cardiopulmonary conditions (acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, or serious ventricular arrhythmias)
* Pregnancy or lactation. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Participants may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Early Tumor Response | Base line up to 24 weeks
  Dynamic CEUS imaging will demonstrate perfusion characteristics that will predict early tumor response to Transarterial Y90 embolization in Hepatocellular Carcinoma. A change in intra-tumoral arterial flow will be predictive of early response. This will be evaluated immediately following hepatic artery embolization (day 0), at 4 weeks (follow-up 1), 12 weeks (follow-up 2) and 24 weeks (follow-up 3). A modified RECIST will be used to measure early tumor response.

SECONDARY OUTCOMES:
Number of Participants with Early Signs of Radiation Induced Liver Disease (RILD) | Base line up to 24 weeks
  Dynamic CEUS imaging will demonstrate perfusion characteristics that will predict early signs of Radiation Induced Liver Disease (RILD) after Transarterial Y90 embolization in Hepatocellular Carcinoma. This will be evaluated immediately following hepatic artery embolization (day 0), at 4 weeks (follow-up 1), 12 weeks (follow-up 2) and 24 weeks (follow-up 3).

CONTACTS AND LOCATIONS:
Overall Officials: Melissa McGettigan, MD, Principal Investigator — Moffitt Cancer Center; Jennifer Sweeney, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided